CLINICAL TRIAL: NCT04273880
Title: Differences by Sex and Genotype in the Effects of Stress on Executive Functions
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adele Diamond, Professor and Tier 1 Canada Research Chair, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H13-00286; 5R01DA037285-05 (NIH)
Record Dates: First submitted 2019-05-27; First posted 2020-02-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stress
MeSH Terms: interventions — Methylphenidate; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10 mg Psychostimulant (Experimental): Drug: Methylphenidate (MPH) Participants will be tested twice, approximately one month apart. In one of the sessions, they will be given 10mg of MPH an hour and a half before the testing session is set to begin, to account for the time taken for the effects of the drug to start.
  Interventions: Drug: Methylphenidate
- 90 mg Vitamin C (Placebo Comparator): Placebo: Vitamin C Participants will be tested twice, approximately one month apart. In one of the sessions, they will be given 90mg of Vitamin an hour and a half before the testing session is set to begin, to follow the exact protocol that is used for MPH.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Methylphenidate — 10mg of MPH taken an hour and a half before one of the testing sessions.
  Other Names: 02249324
  Arms: 10 mg Psychostimulant
Drug: Vitamin C — 90 mg of Vitamin C taken an hour and a half before the other testing session
  Other Names: Ascorbic Acid
  Arms: 90 mg Vitamin C

SUMMARY:
The aim of this project is to test the effects of an environmental factor (mild stress) on prefrontal cortex (PFC) and the cognitive functions that depend on PFC (collectively called executive functions [EFs]), and to test our predictions concerning how those effects differ by biological factors (hormones and genotype). To test our hypotheses concerning mechanism, the investigators will model the effects of mild stress on EFs pharmacologically. The purpose is to pharmacologically model the effects of mild stress on the cognitive functions (collectively called "executive functions" [EFs]) dependent on the frontal lobe. The investigators would also like to investigate how gender differences and genotype mediate the effect of methylphenidate (MPH) on EFs.

DETAILED DESCRIPTION:
The investigators propose to test each young adult twice; once on the lowest clinically relevant dose of MPH and once on a placebo (Vitamin C), with the order counterbalanced. The two testing sessions will be scheduled 4 weeks apart, once 90 minutes after taking 10mg MPH and once 90 minutes after taking a placebo (90 mg of Vitamin C). Peak plasma concentration of MPH is reached approximately 2 h after ingestion, thus to gain the maximum effect of MPH, the investigators will test subjects 90 minutes after ingestion. They will tell subjects that they are studying the effects of low-dose MPH on EFs, and that they expect it to help the EFs of some but hinder those of others, without telling them the study's predictions. Before each testing session, subjects will come to the lab 90 minutes in advance of the testing period. First, they will be given a pill they will take in front of a research assistant (MPH or placebo). The conditions will be counterbalanced across subjects within each subject group. This is a double-blind design, where neither subject nor tester will know which condition they will be in. The pills (10mg MPH, and 90mg Vitamin C) are made to be identical. They will be over-encapsulated with an opaque coloured capsule. The pills will be in kept in sealed containers that are labeled in such a way that neither the subjects, nor the testers, nor the PI, will not know which pill is which, until it is time for the data analysis. Only a pharmacist, at the compounding pharmacy, will know which container contains which pill.

At low doses the mode of action of MPH increases DA efflux specifically in PFC and preferentially enhances signal processing in PFC. Low dosages of MPH are often effective in improving EFs and specifically because of their effect on PFC. This slight increase of DA in the PFC is similar to the effects of mild stress on the brain, which is why the study uses a low dose of MPH as the pharmacological model of mild stress. Even mild stress markedly increases DA levels in PFC, impairing PFC function and EFs. The use of MPH is meant to mimic the effect of mild stress on the PFC and executive functions.

Purpose/objective: This double-blind study aims to compare performance on tasks of executive function between males, females when their estrogen levels are high, and females when their estrogen levels are low when they have undergone a pharmacological model of mild stress (low dosage of MPH) and when they have not undergone this stress. It also aims to compare the same across the three variants of the catechol-O-methyltransferase (COMT) genotype (methionine-methionine, methionine-valine, and valine-valine).

Hypotheses: MPH, like mild-stress, should raise PFC DA levels in COMT-Vals to optimal, but raise PFC DA levels in COMT-Mets past optimal (since low dose of MPH increases DA levels in PFC). While COMT-Mets generally show better EFs than COMT-Vals without MPH, on MPH that should be reversed with COMT-Vals performing better. An increase in PFC DA levels pharmacologically should mimic the sex difference in the effect of mild stress on EFs, harming females with high estrogen level's performance while enhancing males' performance on tasks of executive functions.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 20 and 35 years old

Exclusion Criteria:

* a neurological impairment or disorder, learning disability, or psychological syndrome that might affect EF performance (such as ADHD)
* inability to understand the task instructions (which are in English), or difficulty hearing the instructions, seeing the stimuli, or executing a manual response.
* a serious adverse event during pregnancy or birth.
* an injury (such as a head injury with loss of consciousness) that might affect EF performance.
* a major trauma that might affect current EFs and stress responsivity
* undue current life stress level
* taking any medication that affects thinking, memory, mental clarity, or any other EF ability.
* taking any medication that influences circulating gonadal hormone levels (such as oral contraceptives [birth control pill]).
* having taken such medications within the preceding four months.
* smokers
* use of recreational drugs or consumption of alcohol 24 hours prior to the testing sessions
* women without a period that occurs roughly every month (predicting the onset of the next menses in women who don't have their period monthly is difficult)
* women who are pregnant or who are nursing.
* having the eye problem glaucoma
* having a heart condition
* being anxious, tense or agitated
* taking or have taken within the past 14 days an anti-depression medicine called a monoamine oxidase inhibitor or MAOI.
* taking pressor agents (for hypotension treatment)
* taking coumarin anticoagulants
* taking anticonvulsants (phenobarbital, diphenylhydantoin, primidone)
* taking phenylbutazone (nonsteroidal anti-inflammatory drug)
* taking tricyclic antidepressants (imipramine, desipramine)
* taking cold or allergy medicine that contain decongestants
* being allergic to anything in either the MPH or Vitamin C capsules (methylphenidate HCL, ascorbic acid, lactose, gelatin, Titanium dioxide, D&C Red #28, FD&C Blue #1, FD&C Red #40)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2018-04-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Selective attention as assessed by the Flanker/Reverse Flanker task: Day 1 | Day 1
  In the regular Flanker task, participants must selectively attend to the direction in which the center stimulus is pointing, ignoring the flanking stimuli. They must press the leftmost key or the rightmost key depending on the direction of the center stimulus. In the Reverse Flanker task, participants must selectively attend to the direction in which the flanking stimulus are pointing, ignoring the center stimulus. Response time and accuracy are measured.
Selective attention as assessed by the Flanker/Reverse Flanker task: 1 Month | 1 Month
  In the regular Flanker task, participants must selectively attend to the direction in which the center stimulus is pointing, ignoring the flanking stimuli. They must press the leftmost key or the rightmost key depending on the direction of the center stimulus. In the Reverse Flanker task, participants must selectively attend to the direction in which the flanking stimulus are pointing, ignoring the center stimulus. Response time and accuracy are measured.
Working memory as assessed by the N-back task: Day 1 | Day 1
  In the N-back task, participants must watch a series of letters flash on screen and press the left mouse button whenever the stimulus that appeared was the same as the stimulus that appeared one stimulus prior (e.g. "A, J, A" - press at the second "A"). Response time and accuracy are measured in both tasks.
Working memory as assessed by the N-back task: 1 Month | 1 Month
  In the N-back task, participants must watch a series of letters flash on screen and press the left mouse button whenever the stimulus that appeared was the same as the stimulus that appeared one stimulus prior (e.g. "A, J, A" - press at the second "A"). Response time and accuracy are measured in both tasks.
Working memory as assessed by the Forward Re-Ordering Digit Span task: Day 1 | Day 1
  In the Forward Re-Ordering Digit Span task, participants listen to a series of numbers read out by the tester and they must verbally re-order the numbers in the forward direction. Response time and accuracy are measured in both tasks.
Working memory as assessed by the Forward Re-Ordering Digit Span task: 1 Month | 1 Month
  In the Forward Re-Ordering Digit Span task, participants listen to a series of numbers read out by the tester and they must verbally re-order the numbers in the forward direction. Response time and accuracy are measured in both tasks.
Inhibition as assessed by the Hearts & Flowers task: Day 1 | Day 1
  On the first block of the Hearts & Flowers task, participants must press the button on the same side as a stimulus (e.g. a heart). Then, on the second block, they must press the button on the opposite side as a stimulus (e.g. a flower). Response time and accuracy are measured.
Inhibition as assessed by the Hearts & Flowers task: 1 Month | 1 Month
  On the first block of the Hearts & Flowers task, participants must press the button on the same side as a stimulus (e.g. a heart). Then, on the second block, they must press the button on the opposite side as a stimulus (e.g. a flower). Response time and accuracy are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Diamond, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Developmental Cognitive Neuroscience Lab, Department of Psychiatry, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed at the group level

REFERENCES:
- [Background] Arnsten AF, Goldman-Rakic PS. Noise stress impairs prefrontal cortical cognitive function in monkeys: evidence for a hyperdopaminergic mechanism. Arch Gen Psychiatry. 1998 Apr;55(4):362-8. doi: 10.1001/archpsyc.55.4.362. PMID 9554432
- [Background] Barkley, R. A. (2001). The inattentive type of ADHD as a distinct disorder: What remains to be done. Clinical Psychology: Science and Practice, 8, 489-493.
- [Background] Barkley RA, DuPaul GJ, McMurray MB. Attention deficit disorder with and without hyperactivity: clinical response to three dose levels of methylphenidate. Pediatrics. 1991 Apr;87(4):519-31. PMID 2011430
- [Background] Berridge CW, Devilbiss DM, Andrzejewski ME, Arnsten AF, Kelley AE, Schmeichel B, Hamilton C, Spencer RC. Methylphenidate preferentially increases catecholamine neurotransmission within the prefrontal cortex at low doses that enhance cognitive function. Biol Psychiatry. 2006 Nov 15;60(10):1111-20. doi: 10.1016/j.biopsych.2006.04.022. Epub 2006 Jun 23. PMID 16806100
- [Background] Cerqueira JJ, Mailliet F, Almeida OF, Jay TM, Sousa N. The prefrontal cortex as a key target of the maladaptive response to stress. J Neurosci. 2007 Mar 14;27(11):2781-7. doi: 10.1523/JNEUROSCI.4372-06.2007. PMID 17360899
- [Background] Devilbiss DM, Berridge CW. Cognition-enhancing doses of methylphenidate preferentially increase prefrontal cortex neuronal responsiveness. Biol Psychiatry. 2008 Oct 1;64(7):626-35. doi: 10.1016/j.biopsych.2008.04.037. Epub 2008 Jun 30. PMID 18585681
- [Background] Dickerson SS, Kemeny ME. Acute stressors and cortisol responses: a theoretical integration and synthesis of laboratory research. Psychol Bull. 2004 May;130(3):355-91. doi: 10.1037/0033-2909.130.3.355. PMID 15122924
- [Background] Elliott R, Sahakian BJ, Matthews K, Bannerjea A, Rimmer J, Robbins TW. Effects of methylphenidate on spatial working memory and planning in healthy young adults. Psychopharmacology (Berl). 1997 May;131(2):196-206. doi: 10.1007/s002130050284. PMID 9201809
- [Background] Lataster J, Collip D, Ceccarini J, Haas D, Booij L, van Os J, Pruessner J, Van Laere K, Myin-Germeys I. Psychosocial stress is associated with in vivo dopamine release in human ventromedial prefrontal cortex: a positron emission tomography study using [(1)(8)F]fallypride. Neuroimage. 2011 Oct 15;58(4):1081-9. doi: 10.1016/j.neuroimage.2011.07.030. Epub 2011 Jul 23. PMID 21801840
- [Background] Milich, R., Balentine, A. C., & Lynam, D. R. (2001). ADHD combined type and ADHD predominantly inattentive type are distinct and unrelated disorders. Clinical Psychology: Science and Practice, 8, 463-488.
- [Background] Morrow BA, Roth RH, Elsworth JD. TMT, a predator odor, elevates mesoprefrontal dopamine metabolic activity and disrupts short-term working memory in the rat. Brain Res Bull. 2000 Aug;52(6):519-23. doi: 10.1016/s0361-9230(00)00290-2. PMID 10974491
- [Background] Roth RH, Tam SY, Ida Y, Yang JX, Deutch AY. Stress and the mesocorticolimbic dopamine systems. Ann N Y Acad Sci. 1988;537:138-47. doi: 10.1111/j.1749-6632.1988.tb42102.x. No abstract available. PMID 3059920
- [Background] Schmeichel BE, Zemlan FP, Berridge CW. A selective dopamine reuptake inhibitor improves prefrontal cortex-dependent cognitive function: potential relevance to attention deficit hyperactivity disorder. Neuropharmacology. 2013 Jan;64(1):321-8. doi: 10.1016/j.neuropharm.2012.07.005. Epub 2012 Jul 11. PMID 22796428
- [Background] Spencer RC, Klein RM, Berridge CW. Psychostimulants act within the prefrontal cortex to improve cognitive function. Biol Psychiatry. 2012 Aug 1;72(3):221-7. doi: 10.1016/j.biopsych.2011.12.002. Epub 2011 Dec 29. PMID 22209638
- [Background] Weiss M, Worling D, Wasdell M. A chart review study of the inattentive and combined types of ADHD. J Atten Disord. 2003 Sep;7(1):1-9. doi: 10.1177/108705470300700101. PMID 14738177